CLINICAL TRIAL: NCT04975971
Title: A Retrospective Review of Pain and Inflammation Resolution Outcomes in Patients Who Received DEXTENZA Intracanalicular Dexamethasone (0.4 mg) Insert Prior to or Following Corneal Transplant or Cataract Surgery
Brief Title: A Retrospective Review of DEXTENZA 0.4 mg inseRt Following Corneal Transplant or Cataract Surgery
Status: Completed | Type: Observational
Sponsor: Nicole Fram M.D. (Other)
Responsible Party: Sponsor-Investigator, Nicole Fram M.D., Principal Investigator, Advanced Vision Care
Organization: Advanced Vision Care (Other)
Other Study IDs: AVC-004
Record Dates: First submitted 2021-07-02; First posted 2021-07-26 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Anterior Chamber Inflammation; Ocular Pain; Corneal Edema; Corneal Defect; Penetrating KeratoPlasty; Nuclear Cataract; Cortical Cataract; Cataract Senile
MeSH Terms: conditions — Eye Pain; Corneal Edema | interventions — Calcium Dobesilate; Dexamethasone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dextenza recepient: A Retrospective Review DEXTENZA Intracanalicular Dexamethasone (0.4 mg) Insert Prior to or Following Corneal Transplant or Cataract Surgery
  Interventions: Drug: Dextenza 0.4Mg Ophthalmic Insert

INTERVENTIONS:
Drug: Dextenza 0.4Mg Ophthalmic Insert — DEXTENZA is a corticosteroid intracanalicular insert placed in the punctum, a natural opening in the eye lid, and into the canaliculus and is designed to deliver dexamethasone to the ocular surface for up to 30 days without preservatives.
  Other Names: Dexamethasone 0.4mg

SUMMARY:
A Retrospective Review of Pain and Inflammation Resolution Outcomes in Patients Who Received DEXTENZA Intracanalicular Dexamethasone (0.4 mg) Insert Prior to or Following Corneal transplant or Cataract surgery

DETAILED DESCRIPTION:
A Retrospective Review of Pain and Inflammation Resolution Outcomes in Patients Who Received DEXTENZA Intracanalicular Dexamethasone (0.4 mg) Insert, placed within the lower or upper eye lid canaliculus in conjunction with topical steroid Prior to or Following Corneal transplant or Cataract surgery

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Patients who received DEXTENZA insertion perioperatively.

Exclusion Criteria:

* Any patient who did not receive DEXTENZA insertion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will evaluate n=25 (25 eyes) who underwent corneal transplant or cataract surgery and received DEXTENZA insertion prior to or following surgery as documented in E.H.R
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2021-05-19 (Actual)

PRIMARY OUTCOMES:
Mean change in pain score | Assessed for 3 months after drug insertion
  As measured with the visual analog scale (VAS); between 0 and 100; 0 meaning no pain and 100 meaning worse pain possible
Mean change in inflammation (Cell and Flare) scores | Assessed for 3 months after drug insertion
  As measured by SUN (Standardization on Uveitis Nomenclature) grading scale: absence of cell to be defined as a grade of 0-0.5 and absence of flare to be defined as a grade of: 0-1

SECONDARY OUTCOMES:
Resolution of pain | Assessed for 1 months after drug insertion
  Resolution of pain as assessed by aquestionnaire in post-op visits
Resolution of anterior chamber inflammation | Assessed for 3 months after drug insertion
  Resolution of anterior chamber inflammation as measured by SUN grading at the slitlamp in post-op visits
Proportion of eyes requiring additional post-operative therapy | Assessed for 3 months after drug insertion
  Proportion of eyes requiring additional post-operative therapy for pain and inflammation
Number of patient call-backs regarding post-operative pain | Assessed for 3 months after drug insertion
  Number of patient call-backs regarding post-operative pain and medication management
Number of pharmacy call-backs regarding post-operative medication | Assessed for 3 months after drug insertion
  Number of pharmacy call-backs regarding post-operative medication management
Adverse events | Assessed for 3 months after drug insertion
  Incidence and severity of adverse events
Mean change in IOP | Assessed for 3 months after drug insertion
  Mean change in IOP over post-op visits
Change in BCVA | Assessed for 3 months after drug insertion
  Change in BCVA over post op visits

CONTACTS AND LOCATIONS:
Overall Officials: Nicole R Fram, M.D., Principal Investigator — Advanced Vision Care
Locations (1):
- Advanced Vision Care, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tyson SL, Bafna S, Gira JP, Goldberg DF, Jones JJ, Jones MP, Kim JK, Martel JM, Nordlund ML, Piovanetti-Perez IK, Singh IP, Metzinger JL, Mulani D, Sane S, Talamo JH, Goldstein MH; Dextenza Study Group. Multicenter randomized phase 3 study of a sustained-release intracanalicular dexamethasone insert for treatment of ocular inflammation and pain after cataract surgery. J Cataract Refract Surg. 2019 Feb;45(2):204-212. doi: 10.1016/j.jcrs.2018.09.023. Epub 2018 Oct 24. PMID 30367938
- See also: Dextenza (dexamethasone insert) Prescribing Information, Ocular Therapeutix,Inc.2019 — http://www.dextenza.com/wp-content/uploads/2019/06/NDA-208742-S001-Dextenza-labeling-19Jun19.pdf